CLINICAL TRIAL: NCT01578967
Title: LCCC 1115: A Pilot Feasibility Trial of Induction Chemotherapy With ABVD Followed by Brentuximab Vedotin (SGN-35) Consolidation in Patients With Previously Untreated Non-Bulky Stage I or II Hodgkin Lymphoma (HL)
Brief Title: Induction Chemo w/ABVD Followed by Brentuximab Vedotin Consolidation in Newly Diagnosed, Non-Bulky Stage I/II Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1115
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Hodgkin Lymphoma, Adult
Keywords: Hodgkin's lymphoma; Hodgkin lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABVD followed by Brentuximab vedotin (Other): Single arm trial
  Interventions: Drug: Brentuximab vedotin; Drug: ABVD

INTERVENTIONS:
Drug: Brentuximab vedotin — IV, 1.8mg/kg, every 3 weeks for 6 cycles.
  Other Names: SGN-35; Adcetris
Drug: ABVD — Doxorubicin - 25mg/m2 IV over 3-5 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
  Bleomycin - 10u/m2 IV, Day 1 and 15, every 28 days, 2-6 cycles Vinblastine - 6mg/m2 IV over 3-5 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
  Dacarbazine - 375mg/m2 IV over 30 minutes, Day 1 and 15, every 28 days, 2-6 cycles.

SUMMARY:
The standard chemotherapy for Hodgkin lymphoma is called ABVD which is a combination of 4 chemotherapy drugs (doxorubicin, bleomycin, vinblastine, and dacarbazine). The number of cycles of ABVD chemotherapy Hodgkin lymphoma patients receive is about 4-6 cycles. In addition to the ABVD chemotherapy, patients with Hodgkin lymphoma will routinely receive radiation therapy. The use of chemotherapy and radiation may cause long term treatment related side effects such as heart problems and other cancers. Researchers are trying to find if combining ABVD chemotherapy with new drugs and reducing the number of ABVD chemotherapy cycles given is just as effective as the standard Hodgkin treatment.

Brentuximab vedotin is approved by the United States Food and Drug administration (FDA) for the treatment of Hodgkin lymphoma that has come back (relapsed). For this research study, the use of brentuximab vedotin in newly diagnosed Hodgkin lymphoma is considered investigational. Brentuximab vedotin is an antibody that also has a chemotherapy drug attached to it. Antibodies are proteins that are part of your immune system. They can stick to and attack specific targets on cells. The antibody part of the brentuximab vedotin sticks to a target called cluster of differentiation antigen 30 (CD30). CD30 is an important molecule on some cancer cells and some normal cells of the immune system.

The purpose of this research study is to see the effects of treatment with fewer cycles of the combination chemotherapy, ABVD, followed by the study drug brentuximab vedotin has on study participants and Hodgkins lymphoma.

DETAILED DESCRIPTION:
This study is designed as a single arm pilot feasibility trial using an induction of 2-6 cycles of ABVD (doxorubicin, bleomycin, vinblastine, and dacarbazine) chemotherapy followed by 6 cycles of brentuximab vedotin (SGN-35) consolidation for previously untreated patients with stage I and II non-bulky Hodgkin Lymphoma (HL).

Feasibility will be determined by the percentage of patients who have no clinical evidence of HL, and achieve positron emission tomograph (PET) negative disease post brentuximab consolidation. We anticipate approximately 40 patients will be eligible across participating centers (including UNC, Mayo Clinic, and the UNC Cancer Network (UNCCN)) over a 2 year period. A future phase II study evaluating progression free survival (PFS) after ABVD followed by brentuximab vedotin will be considered feasible if ≥ 13 of 15 patients enrolled in this pilot trial become PET negative after brentuximab vedotin consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated stage I or II non-bulky Hodgkin lymphoma

  * No mediastinal mass >0.33 maximum intrathoracic diameter on chest x-ray (see Appendix B)
  * No adenopathy ≥7.5 cm in its largest diameter
* Measurable disease as assessed by 2 dimensional measurement by CT (>2cm or 1.5 cm if 0.5 cm slices are used, as in spiral CT scan)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Age ≥18 years and ≤60 years of age
* Life expectancy of at least 3 months
* Adequate bone marrow function (without transfusion support within one week of screening) as demonstrated by:

  * Hemoglobin ≥ 8 g/dL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  * Platelet count ≥ 75,000/mm3
* Adequate hepatic and renal function as demonstrated by:

  * Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN)
  * Total serum bilirubin ≤1.5 x ULN
  * Serum creatinine ≤ 2.0 mg/dL
* Negative serum human chorionic gonadotropin (β-hCG) pregnancy test within 72 hours of day 1 of treatment with ABVD in women of child-bearing potential
* Females of childbearing potential, and males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 6 months following the last dose of brentuximab vedotin. Effective contraception is defined as any medically recommended method (or combination of methods) as per standard of care, including abstinence. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy.
* Signed an institutional review board (IRB)-approved informed consent document for this protocol

Prior to Day 1 of brentuximab vedotin, patients must again meet the following inclusion criteria:

* Adequate bone marrow function (without transfusion support within one week of D1 of brentuximab vedotin) as demonstrated by:

  * Hemoglobin ≥ 8 g/dL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  * Platelet count ≥ 75,000/mm3
* Adequate hepatic and renal function as demonstrated by:

  * Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN)
  * Total serum bilirubin ≤1.5 x ULN
  * Serum creatinine ≤ 2.0 mg/dL
* Achieved at least a partial response (PR) (and not progressed) after ABVD therapy

Exclusion Criteria:

* Prior therapies for treatment of HL including involved field radiation therapy or any prior treatment for any malignancy with anthracyclines.
* Bulky disease (defined as a mass measuring > 7.5 cm or one-third the maximal diameter of the thoracic cavity)
* Known central nervous system (CNS) involvement
* Symptomatic pulmonary disease currently requiring regular medication including but not restricted to bronchodilators
* Known history of human immunodeficiency virus (HIV), hepatitis B and hepatitis C (testing is not necessary if patient does not have history of these diseases, and no risk factors for acquisition of these viruses)
* Cardiac disease with left ventricular ejection fraction of less than 45%
* Known hypersensitivity to any excipient contained in the drug formulation of brentuximab vedotin or any component of ABVD
* Medical or other condition that would represent an inappropriate risk to the patient or would likely compromise achievement of the primary study objective
* Other active malignancies with the exception of:

  * Non-melanoma skin cancer
  * Cervical carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
* Pregnant or lactating women

Prior to Day 1 of brentuximab vedotin, please verify the patient does not meet the criteria below:

* Symptomatic pulmonary disease currently requiring regular medication including but not restricted to bronchodilators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-04; Primary Completion 2016-08-10 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Shea, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina at Chapel Hill, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Levine Cancer Istitute, Carolinas Health Care system, Charlotte, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Park SI, Shea TC, Olajide O, Reddy NM, Budde LE, Ghosh N, Deal AM, Noe JF, Ansell SM. ABVD followed by BV consolidation in risk-stratified patients with limited-stage Hodgkin lymphoma. Blood Adv. 2020 Jun 9;4(11):2548-2555. doi: 10.1182/bloodadvances.2020001871. PMID 32516414
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- ABVD Followed by Brentuximab Vedotin: Single arm trial
  Brentuximab vedotin: IV, 1.8mg/kg, every 3 weeks for 6 cycles.
  ABVD: Doxorubicin - 25mg/m2 IV over 3-5 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
  Bleomycin - 10u/m2 IV, Day 1 and 15, every 28 days, 2-6 cycles Vinblastine - 6mg/m2 IV over 3-5 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
  Dacarbazine - 375mg/m2 IV over 30 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
Period: Overall Study
Arm/Group | ABVD Followed by Brentuximab Vedotin
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One patient was not evaluable due to change in diagnosis during ABVD treatment (HL --> gray zone lymphoma).
Arm/Group | ABVD Followed by Brentuximab Vedotin
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 29 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40
Stage [Count of Participants; unit: Participants] — The stage of lymphoma describes the extent of the spread of the tumor, using the terms stage I through IV (1 through 4). Each stage may also be further divided into "A" and "B" categories, based on whether or not the patient is experiencing specific symptoms. Where larger numbers indicate a worse outcome.
  Participants
    I | 2
    IIA | 28
    IIB | 10
Risk [Count of Participants; unit: Participants] — patients with early stage HL can be stratified into two risk groups: Favorable and unfavorable. This is based on the presence or absence of certain clinical features, such as age, B symptoms, erythrocyte sedimentation rate (ESR), large number of regions involved, and large mediastinal adenopathy.
  Participants
    Favorable | 18
    UnFavorable | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Positron Emission Tomography (PET) Negative Disease
Description: Percentage of patients who convert to PET negative disease post consolidation. This is defined by PET with Deauville <=2.
  The Deauville 5-point scoring system is a five-point scoring system for the Fluorodeoxyglucose (FDG) avidity of a Hodgkin's lymphoma or Non-Hodgkin's lymphoma tumor mass as seen on FDG Positron emission tomography:
  Score 1: No uptake above the background Score 2: Uptake ≤ mediastinum Score 3: Uptake > mediastinum but ≤ liver Score 4: Uptake moderately increased compared to the liver at any site Score 5: Uptake markedly increased compared to the liver at any site Score X: New areas of uptake unlikely to be related to lymphoma
Time Frame: 12 months
Population: One patient was not evaluable due to change in diagnosis during ABVD treatment (HL --> gray zone lymphoma). There was one death due to sepsis and hepatic failure, a very rare but known complication of brentuximab vedotin. Leaving 39 evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | ABVD Followed by Brentuximab Vedotin
Number analyzed (Participants) | 39
Participants | 37

2. Secondary Outcome: Number of Participant Who Achieved a Complete Response
Description: Response criteria based on the International Workshop to standardize response criteria for malignant lymphomas. Complete Response is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABVD Followed by Brentuximab Vedotin
Number analyzed (Participants) | 39
Participants | 37

3. Secondary Outcome: Conversion Rate to Complete Response. Number of Participants Who Had a Partial Response Post ABVD Who Converted to a Complete Response.
Description: Conversion rate to Complete Response after brentuximab vedotin in patients with partial response at the end of ABVD therapy. Response criteria based on the International Workshop to standardize response criteria for malignant lymphomas. Complete Response is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. These nodes or masses should be selected according to all of the following: they should be clearly measurable in at least 2 perpendicular dimensions; if possible they should be from disparate regions of the body; and they should include mediastinal and retroperitoneal areas of disease whenever these sites are involved.
Time Frame: 12 months
Population: 4 subjects had a partial response (PR) (Deauville score of 3)
Measure: Count of Participants; unit: Participants
Arm/Group | ABVD Followed by Brentuximab Vedotin
Number analyzed (Participants) | 4
Participants | 3

4. Secondary Outcome: 3 Year Progression Free Survival Rate
Description: Defined as the percentage of participants who did not show relapse/progression or death from any cause occurred at 3 years after the time from ABVD treatment start. Relapse/progression is measured using the Revised Response Criteria for Malignant Lymphoma and is defined as the following: appearance of any new lesion > 1.5 centimeters (cm) in any axis during or at the end of therapy; at least a 50% increase from nadir in the sum of the product of the diameters (SPD) of any previously involved nodes, or in a single involved node, or the size of other lesions; or at least a 50% increase in the longest diameter of any single previously identified node more than 1 cm in its short axis. In addition, lesions should be PET positive if observed in a typical FDG-avid lymphoma or the lesion was positron emission tomography (PET) positive before therapy
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients progression free
Arm/Group | ABVD Followed by Brentuximab Vedotin
Number analyzed (Participants) | 40
percentage of patients progression free | 92 [77 to 97]

5. Secondary Outcome: 3 Year Time to Progression Rate
Description: Defined as the percentage of participants who did not show relapse/progression at 3 years after the time from ABVD treatment start. Relapse/progression is measured using the Revised Response Criteria for Malignant Lymphoma and is defined as the following: appearance of any new lesion > 1.5 centimeters (cm) in any axis during or at the end of therapy; at least a 50% increase from nadir in the sum of the product of the diameters (SPD) of any previously involved nodes, or in a single involved node, or the size of other lesions; or at least a 50% increase in the longest diameter of any single previously identified node more than 1 cm in its short axis. In addition, lesions should be PET positive if observed in a typical FDG-avid lymphoma or the lesion was positron emission tomography (PET) positive before therapy
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients progression free
Arm/Group | ABVD Followed by Brentuximab Vedotin
Number analyzed (Participants) | 40
percentage of patients progression free | 92 [77 to 97]

6. Secondary Outcome: Number of Adverse Events Attributed to Brentuximab Vedotin With a Grade 3 or Higher
Description: Number of adverse events attributed to Brentuximab Vedotin with a grade 3 or higher. Toxicity assessed via the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4. The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.The higher the grade the more severe the adverse event.
Time Frame: 12 months
Population: Please note all grade 4 or higher events were experienced by one patient. The patient developed fever and hepatic dysfunction after 1 dose of Brentuximab Vedotin (BV). Patient also developed pancreatitis and eventually died of sepsis.
Measure: Number; unit: Number of events
Groups:
- Grade 3; Grade 4; Grade 5: Single arm trial
  Brentuximab vedotin: IV, 1.8mg/kg, every 3 weeks for 6 cycles.
  ABVD: Doxorubicin - 25mg/m2 IV over 3-5 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
  Bleomycin - 10u/m2 IV, Day 1 and 15, every 28 days, 2-6 cycles Vinblastine - 6mg/m2 IV over 3-5 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
  Dacarbazine - 375mg/m2 IV over 30 minutes, Day 1 and 15, every 28 days, 2-6 cycles.
Arm/Group | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 40 | 40 | 40
Number of events
  Neutropenia | 3 | 0 | 0
  Infections and infestations | 1 | 0 | 1
  Alanine aminotransferase increased | 1 | 0 | 0
  Anemia | 1 | 0 | 0
  Ascites | 0 | 1 | 0
  Aspartate aminotransferase increased | 1 | 0 | 0
  Blood bilirubin increased | 0 | 1 | 0
  Creatinine increased | 1 | 0 | 0
  Hepatic failure | 0 | 1 | 0
  Hyperglycemia | 1 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0
  Lipase increased | 0 | 1 | 0
  Pancreatitis | 0 | 1 | 0
  Peripheral sensory neuropathy | 1 | 0 | 0
  Platelet count decreased | 0 | 1 | 0
  Pleural effusion | 0 | 1 | 0
  Rash maculo-papular | 1 | 0 | 0
  Renal and urinary disorders | 0 | 1 | 0
  Sepsis | 0 | 0 | 1
  Syncope | 1 | 0 | 0
  White blood cell decreased | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | ABVD Followed by Brentuximab Vedotin
All-Cause Mortality (participants affected / at risk) | 1/41
Serious Adverse Events (participants affected / at risk) | 6/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABVD Followed by Brentuximab Vedotin (N=41)
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Catheter related infection (Infections and infestations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hypotension (Vascular disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 2
Meningitis (Infections and infestations) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ABVD Followed by Brentuximab Vedotin (N=41)
Abdominal Pain (Gastrointestinal disorders) | 2
Alanine Aminotransferase Increased (Investigations) | 18
Alkaline Phosphatase Increased (Investigations) | 6
Allergic Reaction (Immune system disorders) | 2
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 17
Anemia (Blood and lymphatic system disorders) | 24
Anorexia (Metabolism and nutrition disorders) | 11
Anxiety (Psychiatric disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Aspartate Aminotransferase Increased (Investigations) | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Blood And Lymphatic System Disorders - Other, Specify (Blood and lymphatic system disorders) | 3
Blood Bilirubin Increased (Investigations) | 4
Blurred Vision (Eye disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 5
Chills (General disorders) | 9
Constipation (Gastrointestinal disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Creatinine Increased (Investigations) | 3
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 13
Dizziness (Nervous system disorders) | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Edema Limbs (General disorders) | 6
Fatigue (General disorders) | 34
Fever (General disorders) | 9
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 8
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 3
General Disorders And Administration Site Conditions - Other, Specify (General disorders) | 3
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hot Flashes (Vascular disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4/40
Hypoglycemia (Metabolism and nutrition disorders) | 2/40
Hypokalemia (Metabolism and nutrition disorders) | 3/40
Infusion Related Reaction (General disorders) | 2/40
Injection Site Reaction (General disorders) | 3/40
Insomnia (Psychiatric disorders) | 10/40
Lymphocyte Count Decreased (Investigations) | 3/40
Malaise (General disorders) | 9/40
Mucositis Oral (Gastrointestinal disorders) | 7/40
Myalgia (Musculoskeletal and connective tissue disorders) | 8/40
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6/40
Nausea (Gastrointestinal disorders) | 31/40
Neck Pain (Musculoskeletal and connective tissue disorders) | 2/40
Neutrophil Count Decreased (Investigations) | 32/40
Non-Cardiac Chest Pain (General disorders) | 3/40
Pain (General disorders) | 11/40
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5/40
Palpitations (Cardiac disorders) | 2/40
Papulopustular Rash (Infections and infestations) | 2/40
Paresthesia (Nervous system disorders) | 3/40
Peripheral Sensory Neuropathy (Nervous system disorders) | 31/40
Platelet Count Decreased (Investigations) | 3/40
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 3/40
Pruritus (Skin and subcutaneous tissue disorders) | 9/40
Rash Acneiform (Skin and subcutaneous tissue disorders) | 6/40
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 19/40
Sinusitis (Infections and infestations) | 2/40
Skin Infection (Infections and infestations) | 5/40
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4/40
Syncope (Nervous system disorders) | 2/40
Upper Respiratory Infection (Infections and infestations) | 4/40
Urinary Frequency (Renal and urinary disorders) | 2/40
Urinary Tract Pain (Renal and urinary disorders) | 2/40
Urticaria (Skin and subcutaneous tissue disorders) | 2/40
Vomiting (Gastrointestinal disorders) | 10/40
Weight Gain (Investigations) | 5/40
Weight Loss (Investigations) | 2/40
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2/40
White Blood Cell Decreased (Investigations) | 24/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days